CLINICAL TRIAL: NCT00752388
Title: Application of the WHO-5 Well-being Index (WHO-5) as a Screening Instrument for Depression in Parkinson's Disease
Brief Title: Non-interventional Observational Study on WHO-5 Questionnaire Application in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.658
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To assess the predictive value of sequential administration of WHO-5 and MDI (Major Depression Inventory) for the clinical management of Parkinson Disease (PD) patients by

* determination of the prevalence of depression in PD patients, based on MDI severity categories and the self-rating scale WHO-5, where poor well being was indicated.
* exploration of influencing factors (PD status, therapeutic status) on the prevalence of MDI depression categories.

ELIGIBILITY:
Inclusion Criteria:

1. PD patients attending one of the participating neurologist practices during 2 fixed weeks in November 2008
2. Idiopathic PD with or without fluctuations
3. Male or female PD patients aged at least 30
4. Ability to reliably complete self-rating scales (WHO-5, MDI) ), according to the physician's judgement.
5. Written informed consent by the patient for study participation.

Exclusion Criteria:

1. PD Patients who only attend the practice to get a prescription and are not seen by the doctor on that day
2. Patients who are not able to understand the questionnaires (e.g. due to mental impairment or language problems).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: resident physician
Sampling Method: Non-Probability Sample
Enrollment: 1588 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients with depressive symptoms (based on WHO-5 and MDI) in total and in subgroups | day 1

SECONDARY OUTCOMES:
WHO-5 score and items | day 1
MDI score (for a subgroup of patients with WHO-5 score < 13 or any WHO-5 item rated with 0 or 1) | day 1
Correlation of WHO-5 and MDI (for a subgroup of patients with a WHO-5 score < 13 or any WHO-5 item rated with 0 or 1) in PD patients | day 1
Investigator assessment of the applicability of the WHO-5 for screening for depression in PD patients | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (278):
- Germany (278):
  - Boehringer Ingelheim Investigational Site 1, Achim
  - Boehringer Ingelheim Investigational Site 2, Achim
  - Boehringer Ingelheim Investigational Site, Altenburg
  - Boehringer Ingelheim Investigational Site, Altenholz
  - Boehringer Ingelheim Investigational Site, Alzey
  - Boehringer Ingelheim Investigational Site, Aue
  - Boehringer Ingelheim Investigational Site, Bad Driburg
  - Boehringer Ingelheim Investigational Site, Bad Homburg
  - Boehringer Ingelheim Investigational Site, Bad Honnef
  - Boehringer Ingelheim Investigational Site, Bad Neuenahr-Ahrweiler
  - Boehringer Ingelheim Investigational Site 1, Bad Soden
  - Boehringer Ingelheim Investigational Site 2, Bad Soden
  - Boehringer Ingelheim Investigational Site, Bad Sooden-Allendorf
  - Boehringer Ingelheim Investigational Site, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site 10, Berlin
  - Boehringer Ingelheim Investigational Site 11, Berlin
  - Boehringer Ingelheim Investigational Site 12, Berlin
  - Boehringer Ingelheim Investigational Site 13, Berlin
  - Boehringer Ingelheim Investigational Site 14, Berlin
  - Boehringer Ingelheim Investigational Site 1, Berlin
  - Boehringer Ingelheim Investigational Site 2, Berlin
  - Boehringer Ingelheim Investigational Site 3, Berlin
  - Boehringer Ingelheim Investigational Site 4, Berlin
  - Boehringer Ingelheim Investigational Site 5, Berlin
  - Boehringer Ingelheim Investigational Site 6, Berlin
  - Boehringer Ingelheim Investigational Site 7, Berlin
  - Boehringer Ingelheim Investigational Site 8, Berlin
  - Boehringer Ingelheim Investigational Site 9, Berlin
  - Boehringer Ingelheim Investigational Site 1, Bielefeld
  - Boehringer Ingelheim Investigational Site 2, Bielefeld
  - Boehringer Ingelheim Investigational Site 1, Bochum
  - Boehringer Ingelheim Investigational Site 2, Bochum
  - Boehringer Ingelheim Investigational Site 3, Bochum
  - Boehringer Ingelheim Investigational Site, Bockhorn
  - Boehringer Ingelheim Investigational Site, Bonn
  - Boehringer Ingelheim Investigational Site, Braunschweig
  - Boehringer Ingelheim Investigational Site, Bremen
  - Boehringer Ingelheim Investigational Site, Bremerhaven
  - Boehringer Ingelheim Investigational Site, Bretten
  - Boehringer Ingelheim Investigational Site 1, Butzbach
  - Boehringer Ingelheim Investigational Site 2, Butzbach
  - Boehringer Ingelheim Investigational Site, Buxtehude
  - Boehringer Ingelheim Investigational Site, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site, Chemnitz
  - Boehringer Ingelheim Investigational Site, Cloppenburg
  - Boehringer Ingelheim Investigational Site, Coesfeld
  - Boehringer Ingelheim Investigational Site 1, Cologne
  - Boehringer Ingelheim Investigational Site 2, Cologne
  - Boehringer Ingelheim Investigational Site 3, Cologne
  - Boehringer Ingelheim Investigational Site 4, Cologne
  - Boehringer Ingelheim Investigational Site 5, Cologne
  - Boehringer Ingelheim Investigational Site 6, Cologne
  - Boehringer Ingelheim Investigational Site 7, Cologne
  - Boehringer Ingelheim Investigational Site 1, Cottbus
  - Boehringer Ingelheim Investigational Site 2, Cottbus
  - Boehringer Ingelheim Investigational Site, Delmenhorst
  - Boehringer Ingelheim Investigational Site 1, Dessau
  - Boehringer Ingelheim Investigational Site 2, Dessau
  - Boehringer Ingelheim Investigational Site, Dietzenbach
  - Boehringer Ingelheim Investigational Site, Dippoldiswalde
  - Boehringer Ingelheim Investigational Site 1, Dortmund
  - Boehringer Ingelheim Investigational Site 2, Dortmund
  - Boehringer Ingelheim Investigational Site 3, Dortmund
  - Boehringer Ingelheim Investigational Site 1, Dresden
  - Boehringer Ingelheim Investigational Site 2, Dresden
  - Boehringer Ingelheim Investigational Site 3, Dresden
  - Boehringer Ingelheim Investigational Site 4, Dresden
  - Boehringer Ingelheim Investigational Site 1, Duisburg
  - Boehringer Ingelheim Investigational Site 2, Duisburg
  - Boehringer Ingelheim Investigational Site 3, Duisburg
  - Boehringer Ingelheim Investigational Site 4, Duisburg
  - Boehringer Ingelheim Investigational Site, Dülmen
  - Boehringer Ingelheim Investigational Site 1, Düsseldorf
  - Boehringer Ingelheim Investigational Site 2, Düsseldorf
  - Boehringer Ingelheim Investigational Site 3, Düsseldorf
  - Boehringer Ingelheim Investigational Site 4, Düsseldorf
  - Boehringer Ingelheim Investigational Site 5, Düsseldorf
  - Boehringer Ingelheim Investigational Site 1, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site 2, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site, Erftstadt
  - Boehringer Ingelheim Investigational Site, Essen
  - Boehringer Ingelheim Investigational Site 1, Frankfurt
  - Boehringer Ingelheim Investigational Site 2, Frankfurt
  - Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site, Fürstenwalde
  - Boehringer Ingelheim Investigational Site, Gelnhausen
  - Boehringer Ingelheim Investigational Site 1, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 2, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site, Gengenbach
  - Boehringer Ingelheim Investigational Site, Gera
  - Boehringer Ingelheim Investigational Site, Giessen
  - Boehringer Ingelheim Investigational Site, Gifhorn
  - Boehringer Ingelheim Investigational Site, Gladenbach
  - Boehringer Ingelheim Investigational Site, Goch
  - Boehringer Ingelheim Investigational Site, Göttingen
  - Boehringer Ingelheim Investigational Site, Grünstadt
  - Boehringer Ingelheim Investigational Site 1, Güstrow
  - Boehringer Ingelheim Investigational Site 2, Güstrow
  - Boehringer Ingelheim Investigational Site, Gütersloh
  - Boehringer Ingelheim Investigational Site 1, Halle
  - Boehringer Ingelheim Investigational Site 2, Halle
  - Boehringer Ingelheim Investigational Site 3, Halle
  - Boehringer Ingelheim Investigational Site 1, Hamburg
  - Boehringer Ingelheim Investigational Site 2, Hamburg
  - Boehringer Ingelheim Investigational Site 3, Hamburg
  - Boehringer Ingelheim Investigational Site 4, Hamburg
  - Boehringer Ingelheim Investigational Site 5, Hamburg
  - Boehringer Ingelheim Investigational Site, Hamelin
  - Boehringer Ingelheim Investigational Site 1, Hanover
  - Boehringer Ingelheim Investigational Site 2, Hanover
  - Boehringer Ingelheim Investigational Site 3, Hanover
  - Boehringer Ingelheim Investigational Site 4, Hanover
  - Boehringer Ingelheim Investigational Site 1, Heidelberg
  - Boehringer Ingelheim Investigational Site 2, Heidelberg
  - Boehringer Ingelheim Investigational Site, Heilbronn
  - Boehringer Ingelheim Investigational Site, Hemmoor
  - Boehringer Ingelheim Investigational Site, Hennigsdorf
  - Boehringer Ingelheim Investigational Site, Henstedt-Ulzburg
  - Boehringer Ingelheim Investigational Site, Herborn
  - Boehringer Ingelheim Investigational Site, Herzberg
  - Boehringer Ingelheim Investigational Site, Herzogenrath
  - Boehringer Ingelheim Investigational Site 1, Hildesheim
  - Boehringer Ingelheim Investigational Site 2, Hildesheim
  - Boehringer Ingelheim Investigational Site 3, Hildesheim
  - Boehringer Ingelheim Investigational Site 4, Hildesheim
  - Boehringer Ingelheim Investigational Site 5, Hildesheim
  - Boehringer Ingelheim Investigational Site, Homburg
  - Boehringer Ingelheim Investigational Site, Hückelhoven
  - Boehringer Ingelheim Investigational Site, Hürth
  - Boehringer Ingelheim Investigational Site 1, Ilmenau
  - Boehringer Ingelheim Investigational Site 2, Ilmenau
  - Boehringer Ingelheim Investigational Site, Ingelheim
  - Boehringer Ingelheim Investigational Site, Iserlohn
  - Boehringer Ingelheim Investigational Site, Itzehoe
  - Boehringer Ingelheim Investigational Site, Kamen
  - Boehringer Ingelheim Investigational Site, Kamp-Lintfort
  - Boehringer Ingelheim Investigational Site, Kandel
  - Boehringer Ingelheim Investigational Site, Karlstadt am Main
  - Boehringer Ingelheim Investigational Site 1, Kassel
  - Boehringer Ingelheim Investigational Site 2, Kassel
  - Boehringer Ingelheim Investigational Site, Kaufbeuren
  - Boehringer Ingelheim Investigational Site, Kiel
  - Boehringer Ingelheim Investigational Site, Kleinblittersdorf
  - Boehringer Ingelheim Investigational Site, Kleve
  - Boehringer Ingelheim Investigational Site, Lappersdorf
  - Boehringer Ingelheim Investigational Site, Lauterbach
  - Boehringer Ingelheim Investigational Site 1, Leer
  - Boehringer Ingelheim Investigational Site 2, Leer
  - Boehringer Ingelheim Investigational Site 1, Leipzig
  - Boehringer Ingelheim Investigational Site 2, Leipzig
  - Boehringer Ingelheim Investigational Site 3, Leipzig
  - Boehringer Ingelheim Investigational Site 4, Leipzig
  - Boehringer Ingelheim Investigational Site 5, Leipzig
  - Boehringer Ingelheim Investigational Site 1, Leverkusen
  - Boehringer Ingelheim Investigational Site 2, Leverkusen
  - Boehringer Ingelheim Investigational Site, Löbau
  - Boehringer Ingelheim Investigational Site, Ludwigsfelde
  - Boehringer Ingelheim Investigational Site 1, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 2, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 3, Ludwigshafen
  - Boehringer Ingelheim Investigational Site, Ludwigslust
  - Boehringer Ingelheim Investigational Site 1, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 2, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 3, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 4, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 5, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 1, Lüneburg
  - Boehringer Ingelheim Investigational Site 2, Lüneburg
  - Boehringer Ingelheim Investigational Site 1, Lünen
  - Boehringer Ingelheim Investigational Site 2, Lünen
  - Boehringer Ingelheim Investigational Site, Magdeburg
  - Boehringer Ingelheim Investigational Site, Malente
  - Boehringer Ingelheim Investigational Site 1, Mannheim
  - Boehringer Ingelheim Investigational Site 2, Mannheim
  - Boehringer Ingelheim Investigational Site 3, Mannheim
  - Boehringer Ingelheim Investigational Site 4, Mannheim
  - Boehringer Ingelheim Investigational Site, Markkleeberg
  - Boehringer Ingelheim Investigational Site, Marl
  - Boehringer Ingelheim Investigational Site, Memmingen
  - Boehringer Ingelheim Investigational Site, Menden
  - Boehringer Ingelheim Investigational Site, Mittweida
  - Boehringer Ingelheim Investigational Site 1, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 2, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 3, Mönchengladbach
  - Boehringer Ingelheim Investigational Site, Mühlacker
  - Boehringer Ingelheim Investigational Site 1, Mülheim
  - Boehringer Ingelheim Investigational Site 2, Mülheim
  - Boehringer Ingelheim Investigational Site 3, Mülheim
  - Boehringer Ingelheim Investigational Site 1, Münster
  - Boehringer Ingelheim Investigational Site 2, Münster
  - Boehringer Ingelheim Investigational Site 3, Münster
  - Boehringer Ingelheim Investigational Site, Naumburg
  - Boehringer Ingelheim Investigational Site, Neubrandenburg
  - Boehringer Ingelheim Investigational Site, Neuenhagen
  - Boehringer Ingelheim Investigational Site, Neukirchen-Vluyn
  - Boehringer Ingelheim Investigational Site, Neumünster
  - Boehringer Ingelheim Investigational Site, Neustadt
  - Boehringer Ingelheim Investigational Site, Norden
  - Boehringer Ingelheim Investigational Site, Nordhorn
  - Boehringer Ingelheim Investigational Site, Nübel
  - Boehringer Ingelheim Investigational Site, Oberndorf
  - Boehringer Ingelheim Investigational Site, Offenbach
  - Boehringer Ingelheim Investigational Site, Oldenburg
  - Boehringer Ingelheim Investigational Site, Oranienburg
  - Boehringer Ingelheim Investigational Site, Oschatz
  - Boehringer Ingelheim Investigational Site, Osnabrück
  - Boehringer Ingelheim Investigational Site, Paderborn
  - Boehringer Ingelheim Investigational Site, Pirmasens
  - Boehringer Ingelheim Investigational Site, Plauen
  - Boehringer Ingelheim Investigational Site, Potsdam
  - Boehringer Ingelheim Investigational Site, Quakenbrück
  - Boehringer Ingelheim Investigational Site, Rastatt
  - Boehringer Ingelheim Investigational Site, Rathenow
  - Boehringer Ingelheim Investigational Site 1, Regensburg
  - Boehringer Ingelheim Investigational Site 2, Regensburg
  - Boehringer Ingelheim Investigational Site, Remscheid
  - Boehringer Ingelheim Investigational Site, Rendsburg
  - Boehringer Ingelheim Investigational Site, Rheine
  - Boehringer Ingelheim Investigational Site, Ribnitz-Damgarten
  - Boehringer Ingelheim Investigational Site, Riesa
  - Boehringer Ingelheim Investigational Site 1, Rostock
  - Boehringer Ingelheim Investigational Site 2, Rostock
  - Boehringer Ingelheim Investigational Site 3, Rostock
  - Boehringer Ingelheim Investigational Site, Rödermark
  - Boehringer Ingelheim Investigational Site, Rüdersdorf
  - Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site, Salzgitter
  - Boehringer Ingelheim Investigational Site, Schirgiswalde
  - Boehringer Ingelheim Investigational Site, Schleiden
  - Boehringer Ingelheim Investigational Site, Schriesheim
  - Boehringer Ingelheim Investigational Site, Schwelm
  - Boehringer Ingelheim Investigational Site 1, Schwerin
  - Boehringer Ingelheim Investigational Site 2, Schwerin
  - Boehringer Ingelheim Investigational Site, Seeheim-Jugenheim
  - Boehringer Ingelheim Investigational Site, Senftenberg
  - Boehringer Ingelheim Investigational Site 1, Solingen
  - Boehringer Ingelheim Investigational Site 2, Solingen
  - Boehringer Ingelheim Investigational Site 3, Solingen
  - Boehringer Ingelheim Investigational Site, Sömmerda
  - Boehringer Ingelheim Investigational Site 1, Stade
  - Boehringer Ingelheim Investigational Site 2, Stade
  - Boehringer Ingelheim Investigational Site, Stollberg
  - Boehringer Ingelheim Investigational Site 1, Stralsund
  - Boehringer Ingelheim Investigational Site 2, Stralsund
  - Boehringer Ingelheim Investigational Site, Strausberg
  - Boehringer Ingelheim Investigational Site, Telgte
  - Boehringer Ingelheim Investigational Site, Teltow
  - Boehringer Ingelheim Investigational Site, Torgau
  - Boehringer Ingelheim Investigational Site, Trier
  - Boehringer Ingelheim Investigational Site, Troisdorf
  - Boehringer Ingelheim Investigational Site, Vechta
  - Boehringer Ingelheim Investigational Site 1, Velen
  - Boehringer Ingelheim Investigational Site 2, Velen
  - Boehringer Ingelheim Investigational Site 1, Verden an der Aller
  - Boehringer Ingelheim Investigational Site 2, Verden an der Aller
  - Boehringer Ingelheim Investigational Site, Viersen
  - Boehringer Ingelheim Investigational Site, Villingen-Schwenningen
  - Boehringer Ingelheim Investigational Site, Voerde
  - Boehringer Ingelheim Investigational Site 1, Warendorf
  - Boehringer Ingelheim Investigational Site 2, Warendorf
  - Boehringer Ingelheim Investigational Site, Wedel
  - Boehringer Ingelheim Investigational Site, Weida
  - Boehringer Ingelheim Investigational Site, Weil am Rhein
  - Boehringer Ingelheim Investigational Site, Weißenfels
  - Boehringer Ingelheim Investigational Site, Werdau
  - Boehringer Ingelheim Investigational Site, Wesseling
  - Boehringer Ingelheim Investigational Site, Wetzlar
  - Boehringer Ingelheim Investigational Site, Weyhe
  - Boehringer Ingelheim Investigational Site 1, Wismar
  - Boehringer Ingelheim Investigational Site 2, Wismar
  - Boehringer Ingelheim Investigational Site, Wolfratshausen
  - Boehringer Ingelheim Investigational Site, Wolgast
  - Boehringer Ingelheim Investigational Site, Wunstorf
  - Boehringer Ingelheim Investigational Site 1, Wuppertal
  - Boehringer Ingelheim Investigational Site 2, Wuppertal
  - Boehringer Ingelheim Investigational Site, Würzburg
  - Boehringer Ingelheim Investigational Site, Zella-Mehlis
  - Boehringer Ingelheim Investigational Site, Zwickau